CLINICAL TRIAL: NCT07222761
Title: An Open-Label, Randomized Phase 3 Study of Linvoseltamab Monotherapy and Linvoseltamab Plus Carfilzomib Versus Standard of Care Combination Regimens in Patients With Relapsed/Refractory Multiple Myeloma
Brief Title: A Study to Compare Linvoseltamab Monotherapy and Linvoseltamab + Carfilzomib Combination Therapy With Standard-of-Care Combination Regimens in Adult Participants With Relapsed/Refractory Multiple Myeloma (RRMM)
Acronym: LINKER-MM5
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R5458-ONC-2246; 2024-519504-27-00 (EU CTIS Number)
Record Dates: First submitted 2025-10-28; First posted 2025-10-30 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Relapsed and/or Refractory Multiple Myeloma (RRMM)
Keywords: BCMA X CD3 Bispecific Monoclonal Antibody; Bispecific combination therapy; Linvoseltamab; Carfilzomib; Proteasome inhibitor
MeSH Terms: interventions — carfilzomib; daratumumab; Dexamethasone; pomalidomide; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part 1: Arm A (Experimental)
  Interventions: Drug: Linvoseltamab
- Part 1: Arm B (Experimental)
  Interventions: Drug: Linvoseltamab; Drug: Carfilzomib
- Part 2: Arm A (Experimental)
  Interventions: Drug: Linvoseltamab
- Part 2: Arm B (Experimental)
  Interventions: Drug: Linvoseltamab; Drug: Carfilzomib
- Part 2: Arm C (Experimental)
  Interventions: Drug: Carfilzomib; Drug: Daratumumab; Drug: Dexamethasone; Drug: Pomalidomide; Drug: Bortezomib

INTERVENTIONS:
Drug: Linvoseltamab — Administered per the protocol
  Other Names: REGN5458; Lynozyfic™
  Arms: Part 1: Arm A; Part 1: Arm B; Part 2: Arm A; Part 2: Arm B
Drug: Carfilzomib — Administered per the protocol
  Other Names: Kyprolis®
  Arms: Part 1: Arm B; Part 2: Arm B; Part 2: Arm C
Drug: Daratumumab — Administered per the protocol
  Other Names: Darzalex Faspro®; Darzalex®
  Arms: Part 2: Arm C
Drug: Dexamethasone — Administered per the protocol
  Other Names: Dexahexal®
  Arms: Part 2: Arm C
Drug: Pomalidomide — Administered per the protocol
  Other Names: Imnovid®; Pomalyst®
  Arms: Part 2: Arm C
Drug: Bortezomib — Administered per the protocol
  Other Names: Velcade®
  Arms: Part 2: Arm C

SUMMARY:
This study is researching a drug called linvoseltamab (also called "study drug") either given alone or in combination with another anti-myeloma drug called carfilzomib, compared to several standard treatments for progressive Multiple Myeloma (MM) after at least 1 but no more than 3 prior therapies.

The aim of this study is to see if the safety and efficacy of linvoseltamab alone or in combination with carfilzomib can deliver better outcomes (deeper and longer responses that help extend life) than standard treatment options.

The study is looking at several other research questions, including:

* What side effects may happen from taking the study drug
* How much study drug is in the blood at different times
* Whether the body makes antibodies against the study drug (which could make the drug less effective or could lead to side effects)

ELIGIBILITY:
Key Inclusion Criteria:

1. Participant with RRMM who received at least 1 but not more than 3 prior lines of therapy, which must have included treatment with lenalidomide and either a Protease Inhibitor (PI) or anti-CD38 monoclonal antibody
2. Eastern Cooperative Oncology Group (ECOG) performance status score ≤2
3. Confirmed progressive disease according to IMWG criteria during or after the most recent line of therapy

Key Exclusion Criteria:

1. Prior treatment with a T cell-based immunotherapy targeting BCMA, including BCMA-directed bispecific antibodies, Bispecific T-cell Engagers (BiTEs), and Chimeric Antigen Receptor (CAR) T cells. Antibody-drug conjugates targeting BCMA (eg, belantamab mafodotin) are not excluded
2. Diagnosis of plasma cell leukemia, symptomatic amyloidosis (including myeloma-associated amyloidosis), Waldenström macroglobulinemia (lymphoplasmacytic lymphoma), or POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes)
3. Known Central Nervous System (CNS) involvement of myeloma including meningeal involvement
4. History of neurodegenerative condition, Progressive Multifocal Leukoencephalopathy (PML), or CNS movement disorder

NOTE: Other protocol defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 915 (Estimated)
Dates: Start 2026-01-02 (Actual); Primary Completion 2029-06-15 (Estimated); Study Completion 2034-09-17 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Treatment Emergent Adverse Events (TEAEs) | Up to 5 years
  Part 1
Severity of TEAEs | Up to 5 years
  Part 1
Occurrence of Adverse Events of Special Interest (AESI) | Up to 5 years
  Part 1
Severity of AESIs | Up to 5 years
  Part 1
Occurrence of Serious Adverse Events (SAEs) | Up to 5 years
  Part 1
Severity of SAEs | Up to 5 years
  Part 1
Minimal Residual Disease (MRD)-negative Complete Response (CR) | At 12 months
  Part 2
Progression-Free Survival (PFS) per IMWG response criteria as determined by BIRC | Up to 5 years
  Part 2

SECONDARY OUTCOMES:
Occurrence of grade ≥2 Cytokine Release Syndrome (CRS) | Up to 28 days
  Part 1
Timing of grade ≥2 CRS | Up to 28 days
  Part 1
Overall Survival (OS) | Up to 7 years
  Part 2
Achievement of Partial Response (PR) or better per IMWG response criteria as determined by BIRC | Up to 5 years
  Part 2
Achievement of Very Good Partial Response (VGPR) or better per IMWG response criteria as determined by BIRC | Up to 5 years
  Part 2
Achievement of CR or better per IMWG response criteria as determined by BIRC | Up to 5 years
  Part 2
Duration Of Response (DOR) as per IMWG response criteria | Up to 5 years
  Part 2
Time To Progression (TTP) as per IMWG response criteria | Up to 5 years
  Part 2
Time To Next Treatment (TTNT) | Up to 5 years
  Part 2
Second PFS | Up to 5 years
  Part 2
MRD-negative CR criteria at any time | Up to 5 years
  Part 2
Time to PR IMWG response category | Up to 5 years
  Part 2
Time to VGPR IMWG response category | Up to 5 years
  Part 2
Time to CR IMWG response category | Up to 5 years
  Part 2
Time to stringent Complete Response (sCR) IMWG response category | Up to 5 years
  Part 2
Sustained MRD-negative CR | Up to 5 years
  Part 2
Duration of MRD-negative CR | Up to 5 years
  Part 2
Occurrence of TEAEs | Up to 5 years
  Part 2
Severity of TEAEs | Up to 5 years
  Part 2
Occurrence of AESIs | Up to 5 years
  Part 2
Severity of AESIs | Up to 5 years
  Part 2
Occurrence of SAEs | Up to 5 years
  Part 2
Severity of SAEs | Up to 5 years
  Part 2
Concentrations of linvoseltamab in serum over time | Up to 5 years
  Part 2
Incidence of Antidrug Antibodies (ADAs) to linvoseltamab | Up to 5 years
  Part 2
Magnitude of ADAs to linvoseltamab | Up to 5 years
  Part 2
Concentrations total soluble B-cell Maturation Antigen (sBCMA) in serum over time | Up to 5 years
  Part 2
Change from baseline in Global Health Status (GHS)/Quality of Life (QoL), per European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) | Up to 5 years
  Part 2 The EORTC QLQ-C30 is a 30-item validated questionnaire developed to measure patient-reported QoL using 1 GHS/QoL scale, 5 functioning scales (physical, role, emotional, cognitive and social) and 9 symptom scales / items (fatigue, nausea/vomiting, pain, dyspnea, insomnia, appetite loss, constipation, diarrhea and financial difficulties) among patients with cancer.
  Participants rate items on a 4-point scale, with 1 as "not at all" and 4 as "very much."
Change from baseline in Physical Functioning (PF), per EORTC QLQ-C30 | Up to 5 years
  Part 2
Change from baseline in Role Functioning (RF), per EORTC QLQ-C30 | Up to 5 years
  Part 2
Change from baseline in pain, per EORTC QLQ-C30 | Up to 5 years
  Part 2
Change from baseline in fatigue, per EORTC QLQ-C30 | Up to 5 years
  Part 2
Change in patient reported Disease Symptoms (DS) per EORTC Quality of Life Questionnaire-Multiple Myeloma (MM) module 20 [QLQ-MY20]) | Up to 5 years
  Part 2 EORTC QLQ-MY20 is an accompanying 20-item validated questionnaire that measure quality of life among patients living with MM across 4 scales (disease symptoms, side effect of treatment, body image and future perspective). A high score represents a high level of symptoms or problems.
Change in patient reported Treatment Side Effects (TSE) per EORTC QLQ-MY20 | Up to 5 years
  Part 2
Change in patient-reported health state per EuroQoL-5 Dimension-5 Level Scale [EQ-5D-5L]) Visual Analogue Scale (VAS) | Up to 5 years
  Part 2 The EQ-5D-5L is a generic questionnaire that measures HRQoL across 5 dimensions of health (mobility, self-care, usual activities, pain/discomfort and anxiety/depression) across 5 levels (no problems, slight problems, some problems, severe problems and extreme problems) and a VAS of pain (where 0: no pain and 10: worst pain), higher scores indicate higher pain.
Change in patient-reported overall impact of treatment per Functional Assessment of Chronic Illness Therapy (FACIT) item GP5 | Up to 5 years
  Part 2 FACIT Item GP5 is a recommended item by the Federal Drug Administration (FDA) in its recent draft guidance for cancer trials to assess patient-reported overall impact of treatment toxicity. It uses a single item "I am bothered by side effects of treatment" on a 5-point scale (0= not at all, 1= a little bit, 2= somewhat, 3= quite a bit, 4= very much)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (2):
- Gold Coast Hospital and Health Service, Southport, Queensland, Australia
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/